CLINICAL TRIAL: NCT02482402
Title: Iloprost for Bridging to Heart Transplantation in Patients With Pulmonary Hypertension and Left Heart Failure A Randomized, Controlled, Double-blind, Parallel Group, Proof-of-concept Trial
Brief Title: Iloprost for Bridging to Heart Transplantation in PH
Acronym: BRIDGE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Delay in recruitment
Sponsor: Heidelberg University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IG 43; 2013-001613-33 (EudraCT Number)
Record Dates: First submitted 2014-10-31; First posted 2015-06-26 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Chronic Left Ventricular Failure; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Iloprost (Experimental): 2 inhalations per day of 2.5 µg Iloprost [Ventavis®] per inhalation to a maximum of 6 inhalations per day of 5 µg Iloprost per inhalation (total daily dose 5 - 30 µg) will be performed according to each patient's health condition.
  Interventions: Drug: Inhaled Iloprost
- Placebo inhaled (Placebo Comparator): 2 to a maximum of 6 inhalations per day of placebo solution (PLA) will be performed. Study medication will be inhaled using the portable, hand-held I-Neb AAD vibrating mesh technology nebulizer system.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled Iloprost — Treatment effect will be controlled at each study visit and the dose and/or inhalation frequency will be adapted.
  Other Names: Ilomedin
  Arms: Inhaled Iloprost
Drug: Placebo — inhalation solution placebo
  Other Names: inhaled placebo
  Arms: Placebo inhaled

SUMMARY:
Trial Rationale/ Justification To assess efficacy and safety of inhaled Iloprost in treatment naïve patients with left heart failure and pulmonary hypertension, who are on the waiting list for orthotopic heart transplantation. As patients often show increasing hemodynamic values while waiting for a donor organ, the transplantation becomes infeasible at the time of identification of an appropriate donor organ when reaching the exclusion limits. Therefore, there is a high need of improvement and stabilisation of the patients' hemodynamic values as PVR, PAP and TPG. In a retrospective, non-controlled study inhaled Iloprost has already shown a beneficial effect on the hemodynamics as reduction of PVR, TPG and CI (Schulz 2010). Treatment with inhaled Iloprost could stabilize the hemodynamics and prevent the patients from being classified as ineligible by the time an appropriate donor organ is identified.

However, the adverse event profile regarding frequency, time-dependency has to be further validated to show safety and tolerability of inhaled Iloprost in this indication.

All patients can be transferred to a long-term medically supervised observation period with inhaled Iloprost therapy.

DETAILED DESCRIPTION:
Scientific Background In many patients with severe left heart failure (LHF) a chronic pulmonary hypertension (PH) occurs during follow-up leading to a remodeling of pulmonary arteries with an increase in pulmonary artery pressure (PAP), pulmonary vascular resistance (PVR) and transpulmonary gradient (TPG). According to the International Society for Heart and Lung Transplantation and the German Standing Committee on Organ Transplantation, cardiac transplantation is contraindicated if values of PAP, PVR, and/or TPG are above 40 mmHg, 240 dyn x s x cm-5, and 15 mmHg, respectively. Even if the patients show only slightly elevated hemodynamic values at the time of application for transplantation, values most often reach the respective exclusion limits during the waiting period. Patients signed in for transplantation partially are not any longer electable for orthotopic heart transplantation (OHT) at the time of identification of an appropriate donor organ. In the meantime the time on the waiting list for heart transplantation is increasing. In 2001, patients being on the waiting list were undergoing heart transplantation within one year. In contrast, 972 patients were on the waiting list while only 325 heart transplantations were performed in Germany in 2011 (www.eurotransplant.nl).

At present, no specific therapy for PH due to left heart disease is available (Galie 2009), treatment with PAH agents is not recommended due to lack of data (Rosenkranz 2011).

There are only few studies with PH-targeted medication within this indication. Phosphodiesterase inhibitors (e.g. Sildenafil), Endothelin-receptor antagonists and Prostacyclin are potential agents for the treatment of PH during the waiting period for a heart transplantation.

Iloprost is a synthetic analogue of Prostacyclin PGI2. Iloprost dilates systemic and pulmonary arterial vascular beds leading to a reduction of blood pressure.

In a previous study the investigators administered aerosolized Iloprost (ILO) in 14 patients with pulmonary hypertension due to chronic cardiac failure on the waiting list for heart transplantation. Iloprost caused a significant reduction in pulmonary arterial pressure and pulmonary vascular resistance without severe side effects and was more effective than nitric oxide (Sablotzky, Grünig et al. 2002, 2003). In a retrospective non-controlled study in 51 patients awaiting orthotopic heart transplantation Iloprost inhalation caused a significant decrease in PVR (from 458 dyn x s x cm-5 to 345 dyn x s x cm-5), a significant decrease in TPG (21 mmHg to 17 mmHg), and a significant improvement in Cardiac Index (CI) from 2,09 l/min/m2 to 2,23 l/min/m2 (Schulz et al., 2010). In a retrospective non-controlled study low-dose Bosentan improved hemodynamic parameters and 1-year survival rate in 82 end-stage heart failure patients on the waiting list for cardiac transplantation (Hefke et al., 2011).

Randomized-controlled trials are missing within this indication. Sildenafil is not a medication of first choice due to contraindications and as well as many patients waiting for OHT are treated with nitrate (medication due to coronary heart disease). In contrast, inhaled Iloprost has advantageous effects on coronary perfusion. However, in this indication the adverse event profile of inhaled Iloprost regarding frequency and time-dependency is not yet clear. In Germany inhaled Iloprost is administered by the I-Neb AAD-System which allows precise, reproducible dose of the drug.

Due to the positive results in retrospective analyses and in the treatment of patients with pulmonary hypertension, the initiation of this proof-of-concept study seems to be justified.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients of any ethnic origin with left heart insufficiency and secondary PH
* Having fulfilled his/her 18th birthday on Visit 1 (Day -7 to -1) of the study
* Written informed consent (must be available before enrollment in the trial)
* Modified WHO functional class III-IV
* PH diagnosed by right heart catheter showing:

  * Baseline mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg
  * Baseline pulmonary vascular resistance (PVR) > 230 dyn x s x cm-5
  * Baseline transpulmonary gradient (TPG) > 15 mm Hg
* Echocardiogram on Visit 1/Day -7 to -1 consistent with secondary PH, specifically evidence of right ventricular hypertrophy or dilation, and absence of mitral valve stenosis
* Patients receiving maximal conventional left heart failure therapy according to current guidelines (ISHLT Guidelines 2006) including intensified treatment with diuretics and have been stable for at least 2 months before entering the study (i.e. no acute decompensations requiring i.v. diuretic treatment).
* Except for diuretics, vasodilators and antihypertensives, medical treatment should not be expected to change during the entire 12-week study period.
* Negative pregnancy test (β-HCG or urine dipstick) at the start of the trial and appropriate contraception throughout the study for women with child-bearing potential.
* Able to understand and sign the Informed Consent Form
* Ability of subject to understand character and individual consequences of the clinical trial

Exclusion Criteria:

* PH of any cause other than permitted in the entry criteria, e.g. concomitantly to portal hypertension, complex congenital heart disease, reversed shunt, anamestic HIV infection, suspected pulmonary veno-occlusive disease based on pulmonary oedema during a previous vasoreactivity test or on abnormal findings compatible with that diagnosis (septal lines or pulmonary edema detected previously at high resolution computer tomography), congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension
* Contraindication for right heart catheterization
* Severe lung disease: FEV1/FVC <0.5 and total lung capacity < 70% of the normal value
* Any subject who had received any investigational medication within 4 weeks prior to the start of this study or who is scheduled to receive another investigational drug during the course of this study
* Any PAH-specific medication (ERAs, PDE-5-I, Prostacyclins) during the last 30 days prior to inclusion (randomization).
* Known intolerance to inhalation treatment
* Conditions where the effects of inhaled Iloprost on platelets might increase the risk of haemorrhage (e.g. active peptic ulcers, trauma, and intracranial haemorrhage).
* Severe coronary heart disease or unstable angina, myocardial infarction within the last six months
* Cerebrovascular events (e.g. stroke) within the last 3 months
* Active liver disease, porphyria or elevations of serum transaminases >3 x ULN (upper limit of normal) or bilirubin > 1.5 x ULN
* Hemoglobin concentration of less than 75 % of the lower limit of normal
* Systolic blood pressure < 85 mmHg
* History or suspicion of inability to cooperate adequately
* Pregnancy and lactation
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03-17 (Actual); Study Completion 2015-03-17 (Actual)

PRIMARY OUTCOMES:
safety and tolerability measured by adverse events rates | baseline until end of study after 12 weeks
  The primary objective of the clinical trial is to acquire first data on safety and tolerability of inhaled Ilorpost in patients with left heart failure on the waiting list for orthotopic heart transplantation.. This proof-of-concept trial aims to evaluate the safety profile of inhaled Iloprost in this indication.

SECONDARY OUTCOMES:
hemodynamics right atrial pressure | baseline vs. 12 weeks
  Right heart catheterization will be performed at trough level, at least 4 hours after last study drug inhalation, according to 4-8 half-life periods.
hemodynamics pulmonary arterial pressure | baseline vs. 12 weeks
  Right heart catheterization will be performed at trough level, at least 4 hours after last study drug inhalation, according to 4-8 half-life periods.
hemodynamics pulmonary arterial wedge pressure | baseline vs. 12 weeks
  Right heart catheterization will be performed at trough level, at least 4 hours after last study drug inhalation, according to 4-8 half-life periods.
hemodynamics Cardiac output | baseline vs. 12 weeks
  Right heart catheterization will be performed at trough level, at least 4 hours after last study drug inhalation, according to 4-8 half-life periods.
hemodynamics Cardiac index | baseline vs. 12 weeks
  Right heart catheterization will be performed at trough level, at least 4 hours after last study drug inhalation, according to 4-8 half-life periods.
hemodynamics venuous oxygen saturation | baseline vs. 12 weeks
  Right heart catheterization will be performed at trough level, at least 4 hours after last study drug inhalation, according to 4-8 half-life periods.
Echocardiography systolic pulmonary arterial pressure | baseline vs. 12 weeks
Echocardiography Tei index | baseline vs. 12 weeks
Echocardiography right atrial area | baseline vs. 12 weeks
Echocardiography right ventricular area | baseline vs. 12 weeks
Echocardiography tricuspid annular plane systolic excursion | baseline vs. 12 weeks
Echocardiography left ventricular pump function | baseline vs. 12 weeks
WHO functional class | baseline vs. 12 weeks
Lung function tests and Blood Gas analysis | baseline vs. 12 weeks
  Lung function test: Bodyplethysmography (preferred method) including forced vital capacity, forced expiratory volume in one second, FEV1 percent, peak expiratory flow rate, forced expiratory flow, lung volume, diffusion-limited carbon monoxide, Blood gas analysis: capillary or arterial blood gas analysis; partial pressure of oxygen and carbon dioxide, oxygen saturation, supplemental oxygen "yes" or "no" (if the patient receives supplemental oxygen the amount will be recorded in the CRF in litres/minute)
6-minute walking distance and Borg dyspnea Score (CR 10) | baseline vs. 12 weeks
  will be performed according to ATS guidelines. Blood pressure, heart rate and oxygen saturation will be measured before and after the test.
Quality of Life SF 36- questionnaire | baseline vs. 12 weeks
Quality of Life CAMPHOR | baseline vs. 12 weeks
Blood pressure | baseline vs. 12 weeks
  blood pressure and heart rate will be measured after the patient has been at rest for at least 5 minutes.
heart rate measurements | baseline vs. 12 weeks
  blood pressure and heart rate will be measured after the patient has been at rest for at least 5 minutes.
Electrocardiography | baseline to 12 weeks
  For deriving the ECGs the patients should always be in supine position. The ECGs should be derived after a resting period of at least 10 minutes. The investigator will review the ECGs for potential AEs.
Clinical laboratory Haematology | baseline to 12 weeks
Clinical laboratory Leucocytes | baseline to 12 weeks
Clinical laboratory erythrocytes | baseline to 12 weeks
  haemoglobin, haematocrit, platelets Substrates Bilirubin, LDL/HDL, cholesterol, triglycerides, creatinine, uric acid, urea, total protein, albumin, glucose Electrolytes Sodium, potassium, calcium, chloride Enzymes SGOT/ASAT, SGPT/ALAT, Gamma-GT, GLDH, AP, LDH, CK Others INR, PTT, β-HCG test for women with childbearing potential at V1; V5 and V6 Biomarkers CRP, NT-proBNP
Clinical laboratory haemoglobin | baseline to 12 weeks
Clinical laboratory haematocrit | baseline to 12 weeks
Clinical laboratory platelets | baseline to 12 weeks
Clinical laboratory Substrates | baseline to 12 weeks
Clinical laboratory Bilirubin | baseline to 12 weeks
Clinical laboratory LDL/HDL | baseline to 12 weeks
Clinical laboratory cholesterol | baseline to 12 weeks
Clinical laboratory triglycerides | baseline to 12 weeks
Clinical laboratory creatinine | baseline to 12 weeks
Clinical laboratory uric acid | baseline to 12 weeks
Clinical laboratory urea | baseline to 12 weeks
Clinical laboratory total protein | baseline to 12 weeks
Clinical laboratory albumin | baseline to 12 weeks
Clinical laboratory glucose | baseline to 12 weeks
Clinical laboratory Electrolytes | baseline to 12 weeks
Clinical laboratory sodium | baseline to 12 weeks
Clinical laboratory potassium | baseline to 12 weeks
Clinical laboratory calcium | baseline to 12 weeks
Clinical laboratory chloride | baseline to 12 weeks
Clinical laboratory SGOT/ASAT | baseline to 12 weeks
Clinical laboratory SGPT/ALAT | baseline to 12 weeks
Clinical laboratory Gamma-GT | baseline to 12 weeks
Clinical laboratory GLDH | baseline to 12 weeks
Clinical laboratory AP | baseline to 12 weeks
Clinical laboratory LDH | baseline to 12 weeks
Clinical laboratory CK | baseline to 12 weeks
Clinical laboratory INR | baseline to 12 weeks
Clinical laboratory PTT | baseline to 12 weeks
Clinical laboratory β-HCG test for women with childbearing potential at | V1; V5 and V6
Clinical laboratory CRP | baseline to 12 weeks
Clinical laboratory NT-proBNP | baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, MD, Principal Investigator — Thoraxclinic at the University Hospital Heidelberg
Locations (2):
- Germany (2):
  - Klinik für Thorax- und Kardiovaskularchirurgie, Bad Oeynhausen
  - Thoraxclinic at the University of Heidelberg, Heidelberg